CLINICAL TRIAL: NCT04381364
Title: Inhalation of Ciclesonide for Patients With COVID-19: A Randomised Open Treatment Study (HALT COVID-19)
Acronym: HALT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ola Blennow, MD, PhD (Other)
Collaborators: Karolinska University Hospital (Other); Danderyd Hospital (Other); Centrallasarettet Västerås (Other)
Responsible Party: Sponsor-Investigator, Ola Blennow, MD, PhD, Principal Investigator, St Goran's Hospital
Organization: St Goran's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-02183
Record Dates: First submitted 2020-05-07; First posted 2020-05-08 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Covid-19; Pneumonia, Viral; Sars-CoV2
Keywords: Corona virus; Covid-19; Sars-CoV2; Randomized controlled trial; Human; Intervention study; Corticosteroids
MeSH Terms: conditions — COVID-19; Pneumonia, Viral | interventions — ciclesonide

STUDY DESIGN:
Intervention Model Description: This multicenter study is an open-labelled, randomized clinical trial for 1:1 ratio of ciclesonide or control arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medical treatment (Experimental): Treatment with ciclesonide
  Interventions: Drug: Ciclesonide Inhalation Aerosol
- Standard of Care (No Intervention): Standard Medical Care

INTERVENTIONS:
Drug: Ciclesonide Inhalation Aerosol — Ciclesonide 320 µg twice daily for 14 days.
  Other Names: Alvesco
  Arms: Medical treatment

SUMMARY:
Randomized open label clinical trial carried out at study centers in Sweden, including Karolinska University Hospital, S:t Göran Hospital, Danderyd Hospital and Västmanlands Hospital. Patients with COVID-19 who are hospitalized with oxygen therapy are eligible for inclusion. Subjects are randomized to 14 days of inhalation with ciclesonide 360 µg twice daily or to standard of care. Primary outcome is duration of received supplemental oxygen therapy. Key secondary outcome is a composite outcome of death and received invasive mechanical ventilation within 30 days.

ELIGIBILITY:
Inclusion criteria:

* Patients 18 years of age or older who have given their written consent to participate in the study.
* Hospitalized and treated with oxygen for a maximum of 48 hours.
* Verified Covid-19: Positive sample for Sars-Cov2 RNA or a positive Sars-Cov2 antigen test from the upper respiratory tract
* Receives oxygen treatment.
* Negative pregnancy test (women of childbearing potential)
* Willing to exercise contraception categorized as "very effective" according to the Clinical Trial Facilitation Group during ongoing study treatment + 7 days (Appendix 2). (female research participant of childbearing potential)

Exclusion criteria:

* Pregnancy, breast-feeding or planned pregnancy.
* Hypersensitivity to ciclesonide or to any of the excipients.
* Concomitant medication with cortisone, ketoconazole, itraconazole, ritonavir or nelfinavir.
* Treatment with> 8 l oxygen / min or supply of > 50% oxygen with nasal high-flow cannula
* Ongoing palliative care or expected survival of less than 72 hours.
* Expected admission to the intensive care unit within 48 hours.
* Active or inactive pulmonary tuberculosis.
* Severe Liver Failure (Child-Pugh C)
* Diagnosed with pulmonary arterial hypertension (PAH) or fibrosis.
* Mental inability, reluctance or language difficulties that make it difficult to understand the meaning of participating in the study.
* Participates in or has recently participated in a clinical trial in the last 30 days. Previous participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2020-05-29 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Duration of received supplemental oxygen therapy | 30 days after study inclusion
  Time (in days) of received supplemental oxygen therapy (defined as being alive and discharged from hospital to home or at least 48 h of not receiving oxygen therapy during hospitalization).

SECONDARY OUTCOMES:
Invasive mechanical ventilation or all-cause death (key secondary outcome) | 30 days after study inclusion
  Rate of and time to (in days) received invasive mechanical ventilation or all-cause death
All cause death | 30 days after study inclusion
  Rate of and time to (in days) death of any cause
Invasive mechanical ventilation | 30 days after study inclusion
  Rate of and time to (in days) received invasive mechanical ventilation
Remaining dyspnea symptoms | 30-35 days and 5-7 months after inclusion
  Level of remaining dyspnea symptoms according to the Modified Medical Research Council Dyspnea Scale
Need for intensive care | 30 days after study inclusion
  Need for intensive care (yes/no and time to ICU care from inclusion)
Proportion of discharged from the hospital to their home or a nursery home | 30 days after study inclusion
  Proportion of patients who are discharged from the hospital to their home or a nursery home and time to discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel P Andersson, MD, PhD, Principal Investigator — Karolinska University Hospital; Ola Blennow, MD, PhD, Principal Investigator — Capio S:t Görans Hospital and Karolinska University Hospital
Locations (11):
- Sweden (11):
  - Södra Älvsborg hospital, Borås
  - Danderyd Hospital, Danderyd
  - Halmstad hospital, Halmstad
  - Karlskoga Hospital, Karlskoga
  - Örebro University Hospital, Örebro
  - Östersund hospital, Östersund
  - Capio S:t Görans Hospital, Stockholm
  - Karolinska University Hospital Huddinge, Stockholm
  - Växsjö Hospital, Vaxjo
  - Västmanland County Hospital Västerås, Västerås
  - Visby Hospital, Visby

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brodin D, Tornhammar P, Ueda P, Krifors A, Westerlund E, Athlin S, Wojt S, Elvstam O, Neumann A, Elshani A, Giesecke J, Edvardsson-Kallkvist J, Bunpuckdee S, Unge C, Larsson M, Johansson B, Ljungberg J, Lindell J, Hansson J, Blennow O, Andersson DP. Inhaled ciclesonide in adults hospitalised with COVID-19: a randomised controlled open-label trial (HALT COVID-19). BMJ Open. 2023 Feb 22;13(2):e064374. doi: 10.1136/bmjopen-2022-064374. PMID 36813503